CLINICAL TRIAL: NCT06489652
Title: Phase I Clinical Study of in Vivo Distribution and Metabolic Kinetic Characterization of 89Zr-Oxine-RY_SW01 Cell Injection for the Treatment of Systemic Sclerosis
Brief Title: 89Zr-Oxine-RY_SW01 Cell Injection for the Treatment of Systemic Sclerosis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Renocell Biotech Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RYSW202402
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single-dose group (Experimental): 89Zr-Oxine-RY_SW01 Cell Injection 2.0 x 10^6 cells/kg treatment
  Interventions: Drug: 89Zr-Oxine-RY_SW01 Cell Injection

INTERVENTIONS:
Drug: 89Zr-Oxine-RY_SW01 Cell Injection — Biodistribution and metabolic kinetic characterization of zirconium-labeled cells in vivo for the treatment of systemic sclerosis by intravenous infusion of 89Zr-Oxine-RY_SW01 cells injection
  Other Names: RY_SW01 Cell Injection

SUMMARY:
Systemic sclerosis (SSc) tends to progress to involve multiple vital organs within 5 years of diagnosis, significantly impacting patient prognosis and survival. Clinical indications suggest that early intervention is more favorable for long-term outcomes in patients. Although guidelines recommend various drugs for symptomatic treatment, there is currently no standard therapy or effective medication to slow the progression of the disease. Therefore, for patients with diffuse SSc, as defined by a skin score of 10≤mRSS≤30 points, who have been treated with at least two therapies, including steroids, immunosuppressive agents, biologics, etc., within 5 years of diagnosis, the applicant intends to develop a drug that can both modulate the immune system and counteract fibrosis. The goal is to provide long-term benefits to patients through early intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signing of informed consent;
2. Age 18-65 years old (including the threshold), male and female;
3. Diagnosis of SSc according to the 2013 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) diagnostic criteria for systemic sclerosis (SSc);
4. Patients diagnosed with diffuse scleroderma after previous treatment with two or more modalities such as hormones, immunosuppressants, and biologics.

Exclusion Criteria:

1. Percentage of patient's predicted lung function FVC (forceful lung volume) <50% at screening;
2. A previous diagnosis of moderate-to-severe pulmonary hypertension or systolic pulmonary artery pressure >45 mmHg measured by echocardiography at screening;
3. The following conditions existed before the screening: (1) myocardial infarction, stroke, renal crisis, severe intestinal disease, severe hypertension (≥160/100mmHg) uncontrolled patients with the onset or exacerbation of clinical symptoms within 6 months; (2) unstable ischemic heart disease, uncontrolled arrhythmia, cardiac arrhythmia, cardiac tachyarrhythmia, and cardiac tachycardia (≥160/100mmHg) uncontrolled patients with the onset or aggravation of clinical symptoms within 3 months. controlled arrhythmia, heart failure, New York Heart Association stage III/IV or echocardiography suggesting left ventricular ejection fraction <50%, renal insufficiency, renal hypertension, etc;
4. Patients with pre-screening comorbid autoimmune connective tissue diseases other than systemic sclerosis, but with secondary dry syndrome were allowed to participate in this trial;
5. Presence of any of the following laboratory findings at the time of screening:

   ① the presence of abnormal blood routine: hemoglobin <100g / L; white blood cell count <3.0 × 10^9 / L; absolute neutrophil count <1.5 × 10^9 / L; platelet count <100 × 10^9 / L;

   ② abnormal liver function: ALT or AST >3 times the upper limit of normal (ULN); total bilirubin >3 times the ULN; (iii) Abnormal renal function: estimated glomerular filtration rate (eGFR) <60mL/min/1.73m^2 or any uncontrolled clinically significant laboratory test abnormality judged by the investigator to be likely to affect the interpretation of the study data or the subject's participation in the study;
6. Patients with a positive human immunodeficiency virus antibody (anti-HIV-Ab) test, active syphilis, active hepatitis C (hepatitis C antibody positive and HCV-RNA positive), HBsAg positive and HBV-DNA positive during the Screening Period may not be enrolled in the study; and patients with a history of severely active or recurrent bacterial, viral, fungal, parasitic or other infections during the Screening Period ;
7. Live/attenuated vaccination within 2 months prior to enrollment;
8. Any of the following within 3 months prior to enrollment: (i) major trauma or major surgery (including joint surgery), or major surgery required during the study period, which, in the opinion of the investigator, poses an unacceptable risk to the subject; (ii) treatments such as plasma exchange or extracorporeal light replacement; (iii) subjects participating in any other clinical trial;
9. History of any malignancy within 5 years prior to enrollment, except adequately treated or excised basal cell carcinoma of the skin or squamous cell carcinoma of the skin or cervical cancer in situ;
10. Intolerance or contraindication to study treatment, including any of the following:

    (i) Hypersensitivity or allergy to any of the components in the excipients of the product; (ii) No peripheral venous access;
11. Have plans to have children for at least 2 years after injection administration, or are unwilling to use effective contraception with their partner, or have plans for sperm or egg donation;
12. Those who are not suitable for PET/CT, such as those who suffer from claustrophobia;
13. Persons who, in the judgment of the investigator, are not suitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Urine SUV value | 14day
Fecal SUV value | 14day

SECONDARY OUTCOMES:
Modified Rodnan Skin Score (mRSS) | 4、12、24 week
Percentage of FVC projections | 4、12、24 week
Health Assessment Questionnaire Disability Index (HAQ-DI) | 4、12、24 week

IPD SHARING:
Plan to Share IPD: No